CLINICAL TRIAL: NCT03995667
Title: Prophylactic Tumor Treating Fields in Management of Patients With Small Cell Lung Cancer
Brief Title: Tumor Treating Fields (TTFields) Therapy to Manage Brain Metastases in Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: NovoCure Ltd. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Timur Mitin, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00018029; NCI-2020-00574 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018029 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Limited Stage Lung Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prevention (TTFields therapy, questionnaire) (Experimental): Patients undergo TTFields therapy over 18-24 hours daily. Cycles repeat every 4 weeks for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Device: Tumor Treating Fields Therapy

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Device: Tumor Treating Fields Therapy — Optune-Tumor Treating Fields (TTFields). Transducer arrays affixed to scalp, worn continuously.
  Other Names: Alternating Electric Field Therapy; TTF; TTFields

SUMMARY:
This phase II single-arm pilot study will evaluate the safety and preliminary efficacy of Optune-Tumor Treating Fields (TTFields) therapy as a prophylactic approach to reducing small cell lung cancer (SCLC) that has spread to the brain (brain metastases). Optune is a portable battery powered device that produces alternating electrical fields, termed tumor treatment fields ("TTFields") within the human body. These TTFields are applied to the patient by electrically insulated surface transducer arrays, which function to disrupt the rapid cell division of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Observed rate of brain metastases following TTFields therapy at 6 months.

SECONDARY OBJECTIVES:

I. Observed rate of brain metastases following TTFields therapy at 12 months. II. Survival of participants with SCLC after using TTFields therapy. III. Usage and overall safety characteristics of TTFields therapy. IV. Quality of life among participants using TTFields therapy. V. Observed rate of SCLC brain metastases at 6 months from the beginning of the 4th cycle of chemotherapy to development of brain metastases.

OUTLINE:

Participants will receive TTFields therapy on a continuous basis (i.e., 18-24 hours a day, 7 days a week) for a period of 12 months or until the development of brain metastases, whichever comes first. Participants will be able to carry the device in an over-the-shoulder bag or backpack so that they can receive continuous at-home treatment. The investigator or other designated healthcare provider will provide detailed instructions regarding the placement/replacement and positioning of the transducer arrays on the participants head. TTFields are applied to the shaved scalp via two pairs of orthogonally positioned transducer arrays. Each pair of transducer arrays will be centered on the participants shaved head such that one pair is placed on the left and right side of the head, and the second pair placed anteriorly and posteriorly. Transducer arrays should be replaced every 2 to 3 days, with a slight relocation of the new arrays ~2 cm from the prior location.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Pathologically confirmed limited stage (LS)-SCLC or extensive stage (ES)-SCLC

  * LS-SCLC - stage I-III (Tany, Nany, M0) that can be safely treated with radiation doses. Excludes T3-4 due to multiple nodules that are too extensive of have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan
  * ES-SCLC - stage IV (Tany, Nany, M1), or T3-4 due to multiple nodules that are too extensive of have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan
* Must be no more than 6 weeks from having received last dose of chemo- and/or radiotherapy for primary tumor to anticipated start of TTField therapy
* Partial response to standard of care (chemo- and/or radiotherapy) as judged by treating physicians with no evidence of recurrence as observed by thoracoabdominal computed tomography (CT) within 12 weeks of enrollment
* No brain metastases as observed by gadolinium (gd)-magnetic resonance imaging (MRI) within 12 weeks of enrollment
* No previous or currently active second malignancy, with exception of non-metastatic prostate cancer, treated stage I breast cancer, skin malignancies
* Life expectancy of at >= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60)
* Participants must be willing and able to fully comply with the minimum required 18 hours/day of TTField therapy
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

Exclusion Criteria:

* Malignant disease, other than that being treated in this study, with exception of non-metastatic prostate cancer, treated stage I breast cancer, skin malignancies
* Implanted pacemaker, defibrillator or deep brain stimulator, or documented clinically significant arrhythmias
* Active implanted medical device (e.g. deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers, defibrillators, and programmable shunts)

  * External medical devices (e.g., insulin pumps) are permitted
* Skull defect (e.g. missing bone with no replacement)
* Shunt
* Bullet fragments
* Evidence of increased intracranial pressure (midline shift > 5 mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
* Sensitivity to conductive hydrogels
* Pregnant or lactating women
* Underlying serious skin condition on the scalp, which in the opinion of the investigator, would prevent or interfere with TTField therapy
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of participant safety or study results

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timur Mitin, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - OHSU Knight Cancer Institute, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Small Cell Lung Cancer (SCLC) Brain Metastases at 6 Months
Time Frame: 6 months following start of tumor treating fields (TTFields) therapy
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of SCLC Brain Metastases at 12 Months
Time Frame: 12 months following start of TTFields therapy
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival of participants with SCLC after using TTFields therapy. The distribution of overall survival will be graphically described using Kaplan-Meier plot, for all subjects together, and for each disease group (extensive stage and limited stage).
Time Frame: Death or last follow up following start of TTFields therapy, whichever comes first (assessed at 6, 12, 24, 36 and 60 months)
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of TTfield Related Adverse Events
Time Frame: Continuously following start of TTFields therapy (up to 12 months)
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Cognitive Adverse Events (AEs) Using Mini Mental State Exam (MMSE)
Description: Incidence of cognitive AEs will be assessed by measuring changes in MMSE scores over time. Descriptive statistical analysis will be conducted.
Time Frame: Continuously following start of TTFields therapy (up to 12 months)
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Quality of Life Over Time: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30)
Description: Quality of life (QoL) among participants using TTFields therapy evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30). The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). For questions 29 and 30, a 7-points scale is used. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Summary of QoLs and its change over time will be presented graphically.
Time Frame: 6 and 12 months following start of TTFields therapy
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of SCLC Brain Metastases
Time Frame: Up to 180 days from Day 1 of the 4th cycle of chemotherapy (each cycle is 28 days)
Population: Data not collected.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months.
Arm/Group | Prevention (TTFields Therapy, Questionnaire)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (TTFields Therapy, Questionnaire) (N=3)
Dermatitis (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to very low accrual overall, no data was collected for the protocol outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03995667/Prot_SAP_001.pdf